CLINICAL TRIAL: NCT04393948
Title: Pilot Study of Low-Dose Single or Bilateral Whole Lung Irradiation for SARS-CoV-2 Pneumonia
Brief Title: Lung Irradiation for COVID-19 Pneumonia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David E. Kozono, Associate Radiation Oncologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020P001494
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV 2
Keywords: SARS-CoV-2; Radiation Therapy; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- No irradiation (Experimental)
  Interventions: Radiation: Phase 2
- 100 cGy single lung irradiation (Experimental): 100 cGy single lung radiation
  Interventions: Radiation: Phase 1; Radiation: Phase 2
- 100 cGy bilateral lung irradiation (Experimental): 100 cGy bilateral lung radiation
  Interventions: Radiation: Phase 1; Radiation: Phase 2

INTERVENTIONS:
Radiation: Phase 1 — Dose Level 1 - 100 cGy irradiation to a single (right-sided) lung using 6 MV photons delivered using a clinical linear accelerator
  Arms: 100 cGy single lung irradiation
Radiation: Phase 1 — Dose Level 2 - 100 cGy irradiation to both lungs using 6 MV photons delivered using a clinical linear accelerator
  Arms: 100 cGy bilateral lung irradiation
Radiation: Phase 2 — Arm A - No irradiation
  Arms: No irradiation
Radiation: Phase 2 — Arm B - 100 cGy irradiation to a single (right-sided) lung using 6 MV photons delivered using a clinical linear accelerator
  Arms: 100 cGy single lung irradiation
Radiation: Phase 2 — Arm C - 100 cGy irradiation to both lungs using 6 MV photons delivered using a clinical linear accelerator
  Arms: 100 cGy bilateral lung irradiation

SUMMARY:
In this research study the investigators want to learn more about the potential benefit of radiation to the lung to improve the health of patients who are hospitalized with Coronavirus-19 (COVID-19) due to infection with a virus called SARS-CoV-2. This infection causes inflammation of the lung, which can make it difficult to breathe. As a result, patients may need supplemental oxygen or be placed on a ventilator. The investigators believe that low dose radiation therapy to the lung may reduce this inflammation and increase the likelihood that patients will need less oxygen support such as ventilation or supplemental oxygen, or be discharged from the hospital in fewer days, compared to without radiation therapy. The amount of radiation is much lower than what is typically used to treat other conditions such as cancer, although it is higher than the dose used for routine medical imaging.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of SARS-CoV-2 infection by RT-PCR or another approved laboratory test ≤ 3 days before enrollment or ≤ 14 days before enrollment with progressive disease suggestive of ongoing SARS-CoV-2 infection; retesting allowed
* Current hospitalization for ≤ 14 days with SARS-CoV-2 infection at the time of enrollment
* Use of supplemental oxygen or oxygen saturation ≤ 94% on room air
* Age ≥ 40
* May receive antiviral medication (e.g., remdesivir, lopinavir/ritonavir, oseltamivir, favipiravir), antibiotics (e.g., azithromycin), chloroquine, hydroxychloroquine, corticosteroids, statins, anticoagulation, antiplatelet agents (e.g., aspirin) and/or convalescent plasma from recovered individuals off study and/or on study if permitted by the other protocol

Exclusion criteria

* Prior or planned treatment with interleukin inhibitors (e.g., tocilizumab, canakinumab, sarilumab) or TNF-α inhibitors within 14 days of enrollment
* Prior lobectomy or pneumonectomy
* Prior thoracic radiotherapy with cumulative lung V20 > 15% to either lung within 1 year of enrollment, or any radiotherapy resulting in a maximum lung dose of 100 cGy or higher within 14 days of enrollment
* Prior chemotherapy or other systemic therapy with potential for pulmonary toxicity or radiosensitization within 14 days or 5 half-lives, whichever is greater, of enrollment, e.g., bleomycin or gemcitabine
* Prior cancer immunotherapy with an immune checkpoint inhibitor within 60 days of enrollment
* Severe pre-existing heart disease, e.g., New York Heart Association (NYHA) functional class ≥ 3 congestive heart failure
* History of bone marrow or solid organ transplantation
* Known history of autoimmune collagen vascular disease, e.g., scleroderma
* Known hereditary syndrome with increased sensitivity to ionizing radiation, e.g., ataxia-telangiectasia or Fanconi anemia
* Pregnancy
* Inability to be positioned supine and flat for radiation planning and delivery
* Inability to provide informed consent or lack of an authorized representative who can provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Feasibility and safety of treating hospitalized patients with SARS-CoV-2 pneumonia with single or bilateral whole lung irradiation | 4 days after randomization
  Subjects will be treated with 100 cGy irradiation to a single (right-sided) lung (dose level 1) or 100 cGy irradiation to both lungs (dose level 2) following a 3 + 3 dose escalation scheme
Phase 2: Proportion with clinical improvement on a 7-point ordinal scale on day 4 after randomization | 4 days after randomization
  The ordinal scale is an assessment of the clinical status on a given day. Each day, the worst (lowest) score from the previous day will be recorded as the score for that previous day.
  The scale is as follows:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or Extracorporeal Membrane Oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring low flow supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care
  7. Not hospitalized

SECONDARY OUTCOMES:
Improvement or worsening on the 7-point ordinal scale over additional intervals | Up to 30 days after randomization
Rate and duration of use of supplemental oxygen | Up to 30 days after randomization
Rate and duration of fever > 38ºC | Up to 30 days after randomization
Rate and duration of invasive mechanical ventilation | Up to 30 days after randomization
Duration of hospitalization | Up to 30 days after randomization
Proportion of participants with overall survival up to 30 days after randomization | Up to 30 days after randomization
Improvement in radiographic findings related to infection/inflammation; comparisons include on study versus baseline scans and irradiated vs. unirradiated lung in subjects randomized to receive single lung irradiation | Up to 30 days after randomization
Treatment-emergent adverse events | Up to 30 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: David Kozono, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No